CLINICAL TRIAL: NCT00179686
Title: A Multicenter, Single-Arm, Open-Label, Study to Evaluate the Safety and Efficacy of Single-Agent Lenalidomide (Revlimid, CC-5013) in Subjects With Recurrent Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Single-Agent Lenalidomide in Subjects With Recurrent Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NSCL-001
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: celgene; cc-5013; NSCLC; CC5013; Revlimid; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Lenalidomide

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
Subjects who qualify will receive single agent lenalidomide once daily on days 1-21 of 28 day cycles. Subjects will continue until disease progression is documented.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >or = to 18 years at the time of signing the informed consent form
3. Able to adhere to the study visit schedule and other protocol requirements
4. Must have a histologically confirmed diagnosis of non small cell lung cancer that has recurred following at least two prior regimens. Those regimens must have contained both a platinum compound and a taxane either sequentially or in combination
5. Subjects must have measurable disease on cross sectional imaging that is at least 2 cm in the longest diameter.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (see Appendix II).
7. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.

WCBP must agree to have pregnancy tests every 4 weeks while on study drug (every 14 days for women with irregular cycles) and 4 weeks after the last dose of study drug.

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm3 (1.5 x 109/L)
   2. Platelet count <100,000/mm3 (100 x 109/L)
   3. Serum creatinine >2.5 mg/dL (221 mmol/L)
   4. Serum SGOT/AST or SGPT/ALT >5.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. Prior history of malignancies other than non-small cell lung cancer (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for > or = to 1 year.
4. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
5. Pregnant or lactating females.
6. Prior > or = grade 3 allergic reaction/hypersensitivity to thalidomide.
7. Prior > or = grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
8. Prior use of lenalidomide.
9. Use of any standard/experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-03; Study Completion 2006-07

PRIMARY OUTCOMES:
To determine the activity of lenalidiomide in recurrent non-small cell lung cancer. Activity will be assessed by measuring the response rate, tumor control rate, and time to tumor progression.

SECONDARY OUTCOMES:
To evaluate the safety of lenalidomide monotherapy as treatment for subjects with recurrent non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Birmingham Cancer Center, Birmingham, Alabama
  - Rush Cancer Institute, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Cancer and Blood Institute, Metairie, Louisiana
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas